CLINICAL TRIAL: NCT01456390
Title: A Prospective Evaluation of Open-Angle Glaucoma Subjects With One Prior Trabeculectomy Treated Concurrently With One Suprachoroidal Stent and Two Trabecular Micro-bypass Stents and a Postoperative Prostaglandin
Brief Title: Open-Angle Glaucoma Subjects With One Prior Trabeculectomy Treated Concurrently With One Suprachoroidal Stent and Two Trabecular Micro-bypass Stents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-023
Record Dates: First submitted 2011-09-28; First posted 2011-10-20 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle glaucoma; Prior trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iStent and iStent supra (Other): Implantation of two iStent devices and one iStent supra device
  Interventions: Device: iStent and iStent supra

INTERVENTIONS:
Device: iStent and iStent supra — Implantation of two iStent devices and one iStent supra device

SUMMARY:
Evaluation in the eyes of subjects with one prior trabeculectomy on one to three ocular hypotensive medications of the intraocular pressure (IOP) lowering effect of two iStent stents in combination with one iStent supra stent and a postoperative prostaglandin.

DETAILED DESCRIPTION:
Evaluation in the eyes of subjects with one prior trabeculectomy on one to three ocular hypotensive medications of the intraocular pressure (IOP) lowering effect of two iStent stents in combination with one iStent supra stent and a postoperative prostaglandin.

ELIGIBILITY:
Inclusion Criteria:

* Phakic patients or pseudophakic patients with posterior chamber intraocular lenses (PC-IOLs)
* Open-angle glaucoma (including pseudoexfoliative)

Exclusion Criteria:

* Aphakic patients or pseudophakic patients with anterior chamber IOLs (AC-IOLs)
* Prior ALT
* Prior SLT within 90 days of screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Subjects observed at Month 12 who experience a mean medicated diurnal IOP reduction of ≥ 20% vs. baseline mean diurnal IOP | 12 Months
  Primary: Subjects observed at the Month 12 visit who experience a mean diurnal IOP reduction of ≥ 20% vs. baseline mean diurnal IOP, had no glaucoma surgical procedures (incisional or laser surgery prior to the 12 month visit), and no postoperative procedure to reposition or remove the stent prior to the 12 month visit, or additional ocular hypotensive medications within 4 weeks of the Month 12 visit

SECONDARY OUTCOMES:
Mean diurnal IOP < 18mm Hg | 12 months
  Secondary: Subjects observed at the Month 12 visit who experience a mean diurnal IOP < 18 mmHg, had no glaucoma surgical procedures (incisional or laser surgery) prior to the 12 month visit, and no postoperative procedure to reposition or remove the stent prior to the 12 month visit or additional ocular hypotensive medications within 4 weeks of the Month 12 visit

OTHER OUTCOMES:
Safety/adverse event monitoring | 0-61 months
  Rate of ocular adverse events through 61 months
  * Findings from IOP, best corrected visual acuity, visual field, specular microscopy measurements
  * Findings from slit-lamp, fundus and gonioscopic examinations

CONTACTS AND LOCATIONS:
Overall Officials: Lilit A Voskanyan, MD, PhD, Principal Investigator — S.V. Malayan Ophthalmological Center, Yerevan, Armenia
Locations (1):
- S.V. Malayan Ophthalmological Center, Yerevan, Armenia

REFERENCES:
- [Derived] Myers JS, Masood I, Hornbeak DM, Belda JI, Auffarth G, Junemann A, Giamporcaro JE, Martinez-de-la-Casa JM, Ahmed IIK, Voskanyan L, Katz LJ. Prospective Evaluation of Two iStent(R) Trabecular Stents, One iStent Supra(R) Suprachoroidal Stent, and Postoperative Prostaglandin in Refractory Glaucoma: 4-year Outcomes. Adv Ther. 2018 Mar;35(3):395-407. doi: 10.1007/s12325-018-0666-4. Epub 2018 Feb 23. PMID 29476443